CLINICAL TRIAL: NCT01169116
Title: Exclusive Hypofractionated Stereotactic Radiotherapy in Non-resectable Single Brain Metastasis: Prospective Study
Brief Title: Exclusive Hypofractionated Stereotactic Radiotherapy in Non-resectable Single Brain Metastasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3592010
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Cancer; Metastasis
Keywords: radiotherapy; radiation oncology; brain metastasis; metastases; radiosurgery; neurosurgery; hypofractionation; stereotaxy
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: hypofractionated stereotactic radiotherapy — hypofractionated stereotactic radiotherapy with 4 fractions of 7 Gy at the periphery of the brain metastasis with 3 mm margin.

SUMMARY:
Patients with single brain metastasis without other metastatic site have a better prognosis, and they need a better brain metastasis control. For non-resectable and non-radiosurgical brain metastasis, the gold standard treatment is whole-brain irradiation with 30 Gy in 10 fractions, but the local control is not achieved in most of the cases. This study investigate the possibility to increase radiation dose in this metastasis with exclusive hypofractionated stereotactic radiotherapy.

DETAILED DESCRIPTION:
For the planning, patients will undergo magnetic resonance imaging (MRI) 1.5 to 3 Tesla, with contrast and volumetric reconstruction of 1 mm and can be used MRI from the diagnosis of metastasis, if it is compatible with the planning system. Then, there will be individualized mask Mask Set for One Patient 41100 (BrainLAB AG, Heimstetten, Germany) for each patient. Patients will undergo computed tomography (CT) without contrast with 1-mm slices with tracking and stereotactic fixation. The images of MRI and CT are fused in the planning system IPLAN version 4.1 (BrainLAB AG, Heimstetten, Germany), where the plan will be implemented. The clinical target volume (CTV) is the macroscopic disease (GTV) displayed on the sign of T1 contrast. The planning target volume (PTV) is the CTV with 3-mm margin in all directions. Can be used multiple dynamic arcs, static conformal multiple fields, multiple static fields modulated and multiple static arcs. The dose-fractionation scheme will be 4 fractions of 7 Gy at the periphery of the PTV, a once daily on 4 consecutive working days. The dose to the PTV encompassing areas of the brainstem or optic tract will be reduced by 20%. The plans will be standardized at the isocenter. The isodose prescription will be the largest isodose that meets the following criteria: isodose covering at least 95% of the PTV with the prescription dose (V100 ≥ 95%) and 95% of prescription dose covering at least 99% of the PTV (V95 ≥ 99%). The maximum dose should be less than 35 Gy. The dose constraint reported by Ernst-Stecken et al will be respected at the expense of prescription isodose, where the normal brain volume (total brain volume less volume PTV) of 20 cc will not receive a dose of 4 Gy per fraction or larger, there is no maximum size limit of metastasis to be included in the study. Use as an index of compliance reported by the Paddick et al and Radiation Therapy Oncology Group (RTOG). Tests will be done for collision safety tests and quality control to ensure the alignment of isocenters radiation, mechanical and coincidence of lasers (Winston-Lutz test). After all, the patients are treated with 6-MeV photons in the linear accelerator Varian Clinac 600 CD (Varian Medical Systems, Palo Alto, CA, USA) with a system of "micromultileaf" m3 (BrainLAB AG, Heimstetten, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Histopathology of primary tumors: all but the primary characteristics of melanoma cancer, small cell lung cancer, germ cell tumors, leukemia or lymphoma, or primary central nervous system.
* Primary-site: controlled, meaning operated and / or irradiated tumor activity without detectable local
* Meningeal dissemination: none
* Extra-cranial metastases: none
* Pre-irradiation brain: absent
* Number of brain metastases: one
* Location of brain metastasis: brain regions not eligible for surgery (such as the hippocampus, amygdala, motor area, eloquent cortex, thalamus, hypothalamus, basal ganglia, optic tract, midbrain, pons, medulla, corpus callosum and internal capsule) or radiosurgery( metastasis <5 mm from the thalamus, hypothalamus, basal ganglia, optic tract, midbrain, pons, medulla, corpus callosum and internal capsule, and / or ≥ 10 ml or ≥ 3 cm in greatest diameter, or 10 ml tissue receiving ≥ 12 Gy).
* Karnofsky Performance Status ≥ 70%
* Informed consent: authorized

Exclusion Criteria:

* patients that don't have the eligibility below

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
feasibility | 1 year
  Through this study we prospectively evaluate the alternative of performing exclusive hypofractionated stereotactic radiotherapy for patients with single brain metastasis that is not eligible for surgery or radiosurgery, with a good prognosis for survival and lower risk of metachronous brain metastases, the primary objective being to verify whether the treatment is feasible in clinical practice.

SECONDARY OUTCOMES:
survival | 1 year
  As a secondary objective, we will evaluate local control, tumor reduction, quality of life, overall survival, whole-brain irradiation free survival and acute and late toxicities related to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Nakamura, MD, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil